Open-label pilot to test a novel 1 Hz intensive repetitive transcranial magnetic stimulation paradigm in patients with anxiety.

Principal Investigator Nicholas Balderston

**NIH Grant Number** 

**IRB Number:** 850766

ClinicalTrials.gov Number NCT05306977

**Current version** 02/14/2022 V - 0.1 **Previous Versions** 

**Study Summary** 

Title

Open-label pilot to test a novel 1 Hz intensive repetitive

transcranial magnetic stimulation paradigm in patients with

anxiety.

**Short Title** Open-label 1 Hz rTMS pilot

**IRB Number** 

Phase Pilot Study

Methodology Open-label

Study Duration 1 years

Study Center(s) Single-center

Aim 1: Determine the effect of a 1-week course of intensive 1

Hz stimulation on anxiety potentiated startle

**Objectives** 

Aim 2: Determine the effect of a 1-week course of intensive 1

Hz stimulation on attention control.

Number of Subjects

10

Main Inclusion and Exclusion Criteria

Anxiety patients, between 18 – 50 years old, free of psychological and neurological conditions, free of contra-

indications for TMS and MRI

**Aim 1:** Outcome measures. Anxiety potentiated startle (APS) Statistical Analysis. The main analysis will be a paired-sample t-test (pre vs. post stimulation).

## Statistical Methodology

**Aim 2:** Outcome measures. Accuracy and reaction time during the visual short term memory task (VSTM). Statistical Analysis. The main analysis will be a 2 [stimulation: pre-stimulation vs. post-stimulation] by 2 [load: low vs. high] repeated-measures ANOVA.

## Data and Safety Monitoring Plan

The Principal Investigator is responsible for detecting, documenting, and reporting unanticipated problems (UPs), adverse events (AEs), including serious adverse events (SAEs), and deviations in accordance with IRB requirements and federal regulations.